CLINICAL TRIAL: NCT01095328
Title: Cost-effectiveness of a Screening Strategy for Q Fever Among Pregnant Women in Risk Areas: a Clustered Randomized Controlled Trial
Brief Title: A Screening Strategy for Q Fever Among Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Dr. E. Hak, Epidemiology, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NL30340.042.09
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-02

CONDITIONS: Q Fever
Keywords: Q fever; Pregnancy; Screening; Cost-effectiveness
MeSH Terms: conditions — Q Fever | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Screening for Q-fever during pregnancy
  Interventions: Other: screening
- control (No Intervention): No screening for Q-fever during pregnancy
  Interventions: Other: screening

INTERVENTIONS:
Other: screening — screening for Q-fever with a single blood sampling

SUMMARY:
Q fever in the Netherlands is becoming more common. A Q fever infection is a serious threat to certain risk groups,including pregnant women. Pregnant women are more often than the general population asymptomatic. Studies from France show that an infection with Coxiella burnetii may cause obstetric complications including spontaneous abortion, intrauterine fetal death, intrauterine growth retardation and oligohydramnios.

The aim of this study is to assess the effectiveness and cost effectiveness of a multidisciplinary screening program, whereby pregnant women in first line healthcare in high-risk areas for Q fever are screened with a single blood sample during pregnancy. If found positive for Q fever, advise for antibiotic treatment will follow as part of regular healthcare. Treatment is therefore not part of the study protocol.

The results of this study will give more insights in the risks of asymptomatic Q fever in pregnancy and the benefits and harms of a screening strategy during pregnancy. This study will be used to give an evidence based advice to the Dutch minister of health on screening for Q fever in pregnancy.

DETAILED DESCRIPTION:
We will conduct a clustered randomized controlled trial among pregnant women within an area of high transmission. The study participants will be recruited by the midwives in high risk areas, defined by postal code from the RIVM. To inform the public in this area about the study we will publish an article in local newspapers. The midwife centers will be randomized to recruit pregnant women for either the control group or the intervention group. The pregnant women will receive study information by mail using the midwives patients file. It is estimated that approximately 10,000 eligible women live in the areas of transmission. After written informed consent, they will start with the strategy for which the midwife center is randomized.

Participants will be asked for a blood sample in their second trimester of pregnancy, possibly combined with the routine structural ultrasound around 20 weeks of pregnancy to minimize hospital visit. If participants are enrolled in their third trimester, they will have their blood sampling as soon as possible after inclusion.

When taking part in the intervention group the sample will be tested immediately for Q fever. If found positive for acute or chronic Q fever, patients have to be referred, according to local protocol, to a hospital for further pregnancy monitoring and long-term bacteriostatic treatment. Follow-up blood samples are required at 14 days, 3, 6 and 12 months after the first blood sampling as part of the standardized control of Q fever disease to diagnose possible chronicity of infection. Furthermore, current routine for pregnant women being treated with antibiotics against Q fever is to perform monthly blood analyses to monitor treatment, and if the serological parameters descend, these controls are brought back to once every two months. According to local protocol patients with Q fever have to deliver in hospital. After pregnancy serology should be continued with check-ups at 3, 6 and 12 months following the current protocol. Furthermore, after delivery a bacteriocide treatment with doxycycline or an alternative will be started by the specialist as part of regular health care.

In the control arm the blood samples will be stored, and analyzed for Q fever after delivery. If tested positive for Q fever after pregnancy antibiotics could be started if needed as part of regular health care.

At baseline, a questionnaire will be administered to all participants asking about the current pregnancy , pregnancy outcome of any previous pregnancies and demographics. Further risk factors for pregnancy outcome will also be obtained such as smoking and drinking behavior, risk-elevating comorbidities and medication use.

After delivery all relevant outcome data will be collected by questionnaires filled out by the midwife, GP or specialist after delivery, notably the presence of obstetric complications. One month after delivery or end of pregnancy, a last questionnaire will be administered to the participant to verify potential long-term consequences of Q fever, potential loss of income, health-related quality-of-life, fatigue and depressive symptoms. Furthermore questions will be asked about the condition of the newborn and risk-accessing questions for Q fever infection will be asked.

In the context of the secondary research questions an extra blood sample will be required, and placentas as well as amniotic fluid will be collected after delivery. The latter will only take place in a limited number of women and only if they gave birth in a hospital.

All participants will receive usual care and will be asked to visit the general practitioner if symptoms of Q fever occur. He/she will start diagnostic research and treatment or will refer the patient to the hospital. Furthermore, both arms have access to an expert team for support.

ELIGIBILITY:
Inclusion Criteria:

* being pregnant under first line healthcare
* being eighteen years or older
* having signed an informed consent form
* having a estimated date of delivery between June 1th 2010 en December 31th 2010

Exclusion Criteria:

* unable to fulfill study procedures
* absence of informed consent
* have been tested positive for Q fever prior to pregnancy
* unable to understand Dutch

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-02 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
obstetric or maternal complications in Q fever positive women | obstetric complications till delivery, maternal till one month post partum
  Presence of any obstetric or maternal complication after the first trimester of pregnancy, i.e. spontaneous abortion, intrauterine fetal death, termination of pregnancy, oligohydramnios, premature delivery or intrauterine growth retardation. Spontaneous abortion is defined as spontaneous expulsion of the embryo or the fetus before 16 weeks of gestation. Oligohydramnios is defined as the ultrasonic measurement with an amniotic index <=5 cm. IUGR is defined as a fetal birth weight less than the 10th percentile for gestational age, according to the national reference curves.

SECONDARY OUTCOMES:
course of infection in pregnant women | till one month post partum
  maternal chronic infection or reactivation
the accuracy of the diagnostic tests used for screening | around 20 weeks of gestation
  the accuracy of the diagnostic tests used for screening (serology vs PCR)
placentitis | one month post partum
  the extent to which the placenta has been infected
costs | till one month post partum
  The costs associated with health care consumption and other related costs among pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Eelko Hak, Dr., Study Director — University Medical Center Groningen; Janna Munster, MD, MSc, Principal Investigator — University Medical Center Groningen; Wim van der Hoek, Drs., Principal Investigator — Center for Infectious Disease Control; Ronald Stolk, Prof. dr., Study Chair — University Medical Center Groningen; Jan Aarnoudse, Prof. dr., Principal Investigator — University Medical Center Groningen; Sander Leenders, Dr., Principal Investigator — Jeroen Bosch Hospital; Bert Timmer, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Background] Hartzell JD, Wood-Morris RN, Martinez LJ, Trotta RF. Q fever: epidemiology, diagnosis, and treatment. Mayo Clin Proc. 2008 May;83(5):574-9. doi: 10.4065/83.5.574. PMID 18452690
- [Background] Carcopino X, Raoult D, Bretelle F, Boubli L, Stein A. Managing Q fever during pregnancy: the benefits of long-term cotrimoxazole therapy. Clin Infect Dis. 2007 Sep 1;45(5):548-55. doi: 10.1086/520661. Epub 2007 Jul 17. PMID 17682987
- [Background] Parker NR, Barralet JH, Bell AM. Q fever. Lancet. 2006 Feb 25;367(9511):679-88. doi: 10.1016/S0140-6736(06)68266-4. PMID 16503466
- [Background] Schimmer B, Morroy G, Dijkstra F, Schneeberger PM, Weers-Pothoff G, Timen A, Wijkmans C, van der Hoek W. Large ongoing Q fever outbreak in the south of The Netherlands, 2008. Euro Surveill. 2008 Jul 31;13(31):18939. No abstract available. PMID 18761906
- [Background] Karagiannis I, Morroy G, Rietveld A, Horrevorts AM, Hamans M, Francken P, Schimmer B. Q fever outbreak in the Netherlands: a preliminary report. Euro Surveill. 2007 Aug 9;12(8):E070809.2. doi: 10.2807/esw.12.32.03247-en. No abstract available. PMID 17868551
- [Background] Van Steenbergen JE, Morroy G, Groot CA, Ruikes FG, Marcelis JH, Speelman P. [An outbreak of Q fever in The Netherlands--possible link to goats]. Ned Tijdschr Geneeskd. 2007 Sep 8;151(36):1998-2003. Dutch. PMID 17953175
- [Background] Jover-Diaz F, Robert-Gates J, Andreu-Gimenez L, Merino-Sanchez J. Q fever during pregnancy: an emerging cause of prematurity and abortion. Infect Dis Obstet Gynecol. 2001;9(1):47-9. doi: 10.1155/S1064744901000084. PMID 11368259
- [Background] Lin JM, Brimmer DJ, Maloney EM, Nyarko E, Belue R, Reeves WC. Further validation of the Multidimensional Fatigue Inventory in a US adult population sample. Popul Health Metr. 2009 Dec 15;7:18. doi: 10.1186/1478-7954-7-18. PMID 20003524
- [Background] Maurin M, Raoult D. Q fever. Clin Microbiol Rev. 1999 Oct;12(4):518-53. doi: 10.1128/CMR.12.4.518. PMID 10515901
- [Background] Langley JM, Marrie TJ, Leblanc JC, Almudevar A, Resch L, Raoult D. Coxiella burnetii seropositivity in parturient women is associated with adverse pregnancy outcomes. Am J Obstet Gynecol. 2003 Jul;189(1):228-32. doi: 10.1067/mob.2003.448. PMID 12861167
- [Background] Raoult D, Fenollar F, Stein A. Q fever during pregnancy: diagnosis, treatment, and follow-up. Arch Intern Med. 2002 Mar 25;162(6):701-4. doi: 10.1001/archinte.162.6.701. PMID 11911725
- [Background] Advice Dutch Health Council, http://www.gezondheidsraad.nl/nl/adviezen/briefadviesbijeenkomst- over-q-koorts-nederland
- [Background] Vaidya VM, Malik SV, Kaur S, Kumar S, Barbuddhe SB. Comparison of PCR, immunofluorescence assay, and pathogen isolation for diagnosis of q fever in humans with spontaneous abortions. J Clin Microbiol. 2008 Jun;46(6):2038-44. doi: 10.1128/JCM.01874-07. Epub 2008 Apr 30. PMID 18448698
- [Background] Wagner-Wiening C, Brockmann S, Kimmig P. Serological diagnosis and follow-up of asymptomatic and acute Q fever infections. Int J Med Microbiol. 2006 May;296 Suppl 40:294-6. doi: 10.1016/j.ijmm.2006.01.045. Epub 2006 Mar 9. PMID 16524773
- [Background] Gikas A, Kofteridis DP, Manios A, Pediaditis J, Tselentis Y. Newer macrolides as empiric treatment for acute Q fever infection. Antimicrob Agents Chemother. 2001 Dec;45(12):3644-6. doi: 10.1128/AAC.45.12.3644-3646.2001. PMID 11709360
- [Background] Stein A, Raoult D. Q fever during pregnancy: a public health problem in southern France. Clin Infect Dis. 1998 Sep;27(3):592-6. doi: 10.1086/514698. PMID 9770161
- [Background] McCaughey C, McKenna J, McKenna C, Coyle PV, O'Neill HJ, Wyatt DE, Smyth B, Murray LJ. Human seroprevalence to Coxiella burnetii (Q fever) in Northern Ireland. Zoonoses Public Health. 2008 May;55(4):189-94. doi: 10.1111/j.1863-2378.2008.01109.x. PMID 18387140
- [Background] Meekelenkamp JCE, Notermans DW, Rietveld A, Marcelis JH, Schimmer B, Reimerink JHJ, Vollebergh JHA, Wijkmans CJ, Leenders ACAP. Seroprevalence of Coxiella burnetii in pregnant women in the province of Noord-Brabant in 2007. Infectieziekten Bulletin, 20: 57-61 [in Dutch].
- [Background] Dupont HT, Thirion X, Raoult D. Q fever serology: cutoff determination for microimmunofluorescence. Clin Diagn Lab Immunol. 1994 Mar;1(2):189-96. doi: 10.1128/cdli.1.2.189-196.1994. PMID 7496944
- [Derived] Munster JM, Leenders AC, Hamilton CJ, Meekelenkamp JC, Schneeberger PM, van der Hoek W, Rietveld A, de Vries E, Stolk RP, Aarnoudse JG, Hak E. Routine screening for Coxiella burnetii infection during pregnancy: a clustered randomised controlled trial during an outbreak, the Netherlands, 2010. Euro Surveill. 2013 Jun 13;18(24):20504. PMID 23787163
- [Derived] Munster JM, Leenders AC, van der Hoek W, Schneeberger PM, Rietveld A, Riphagen-Dalhuisen J, Stolk RP, Hamilton CJ, de Vries E, Meekelenkamp J, Lo-Ten-Foe JR, Timmer A, De Jong-van den Berg LT, Aarnoudse JG, Hak E. Cost-effectiveness of a screening strategy for Q fever among pregnant women in risk areas: a clustered randomized controlled trial. BMC Womens Health. 2010 Nov 1;10:32. doi: 10.1186/1472-6874-10-32. PMID 21040534